CLINICAL TRIAL: NCT04478292
Title: A Phase 3 Multi-institutional Study for Treatment of Children With Newly Diagnosed Hepatoblastoma Using a Modified PHITT Strategy Incorporating a Randomized Assessment of Sodium Thiosulfate as Otoprotection for Children With Localized Disease, and Response Adapted Therapy for Patients With Metastatic Disease
Brief Title: A Multi-institutional Study for Treatment of Children With Newly Diagnosed Hepatoblastoma Using a Modified PHITT Strategy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCMC-SH-HEP-2020
Record Dates: First submitted 2020-06-08; First posted 2020-07-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hepatoblastoma
Keywords: hepatoblastoma, sodium thiosulfate, auditory protection
MeSH Terms: conditions — Hepatoblastoma | interventions — sodium thiosulfate; Cisplatin; Fluorouracil; Vincristine; Biopsy; Transplantation; Doxorubicin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): * Group A1： tumor is completely resected at diagnosis and receives no adjuvant chemotherapy（well differentiated fetal [WDF] histology HB) ；
  * Group A2：tumor is completely resected followed by 2 cycles of standard dose cisplatin monotherapy （non-well differentiated fetal histology HB)
  Interventions: Procedure: Primary surgery resection; Drug: mono CDDP-Group A2
- Group B (Experimental): * Patients will be randomized to one of 2 arms: Arm CDDP or Arm CDDP plus STS. In each arm, patients will be stratified by resectablity after completion of 2 cycles of protocol therapy (6 cycles of standard dose cisplatin monotherapy with or without STS). All the patients in 2 arms will receive 6 cycles chemotherapy in total.
  * Resection of the primary tumor will be performed after completing the 2nd cycle of chemotherapy.
  * Those patients whose tumors after 2 cycles do not meet criteria for definitive surgical, 2nd resectablity evaluation will be scheduled after 4 cycles of chemotherapy.
  Interventions: Drug: Sodium Thiosulfate Injection; Procedure: Biopsy; Procedure: Resection or transplant; Drug: mono CDDP- Group B
- Group C (Experimental): * Patients in Group C will have locally advanced tumors including PRETEXT I-III tumors with a positive VPEFR annotation factor and all PRETEXT IV tumors.
  * Patients will be randomized to one of 2 arms: Arm C5VD or Arm C5VD plus STS. In each arm, patients will be stratified by resectablity after completion of 2 cycles of protocol therapy. All the patients in 2 arms will receive 6 cycles chemotherapy in total.
  * Resection of the primary tumor will be performed after completing the 2nd cycle of chemotherapy.
  * Those patients whose tumors after 2 cycles do not meet criteria for definitive surgical, 2nd resectablity evaluation will be scheduled after 4 cycles of chemotherapy.
  Interventions: Drug: Sodium Thiosulfate Injection; Drug: Cisplatin, 5-Fluorouracil, Vincristine, Doxorubicin-Group C; Procedure: Biopsy; Procedure: Resection or transplant
- Group D (Experimental): * These patients have metastatic disease, suspected HB patients ≥ 8 years of age, or have an AFP ≤ 100 at diagnosis.
  * Patients will receive initial chemotherapy according to the cisplatin-intensive SIOPEL-4 induction regimen. Resection (including transplant) of the primary tumor should be completed after induction Block 3, but primary tumor resection can be planned any time after completing induction therapy.
  * Following 3 blocks of induction chemotherapy, patients will be stratified into 2 risk groups: Group D1 includes patients who either have a chemotherapy-induced lung CR or are rendered a lung CR by surgical metastasectomy. These patients will have chemotherapy consolidation with carboplatin/doxorubicin. In Group D2, patients will have not yet achieved a lung CR at the end of induction Block 3. These patients will get intensified consolidation therapy of carboplatin/doxorubicin with vincristine/irinotecan.
  * Resection of pulmonary nodules should be considered in Group D2.
  Interventions: Procedure: Biopsy; Procedure: Resection or transplant; Procedure: Resection of pulmonary nodules; Drug: Block 1 to 3 (Cisplatin, Doxorubicin) Group D; Drug: Consolidation (Carboplatin, Doxorubicin) -Group D1; Drug: Consolidation (Carboplatin +Doxorubicin/Vincristine + Irinotecan)-Group D2

INTERVENTIONS:
Drug: Sodium Thiosulfate Injection — Weight ≥ 10 kg: 20 g/m2/dose STS or Weight 5-10 kg: 15 g/m2/dose STS or Weight < 5 kg: 10 g/m2/dose STS will be administered by IV over 2 hours beginning 6 hours after the completion of each cisplatin infusion.
  Other Names: STS
  Arms: Group B; Group C
Procedure: Primary surgery resection — Resection of the primary tumor up-front
  Arms: Group A
Drug: mono CDDP-Group A2 — Cisplatin 100 mg/m2/dose Day 1 . All non-WDF patients (A2) will receive 2 cycles of mono cisplatin (100 mg/m2/dose) chemotherapy. Each cycle lasts 3 weeks (21 days).
  Arms: Group A
Drug: Cisplatin, 5-Fluorouracil, Vincristine, Doxorubicin-Group C — All the patients in Group C (2 arms) will receive 6 cycles chemotherapy in total. Cisplatin 100 mg/m2/dose Day 1; 5-Fluorouracil 600 mg/m2/dose Day 1; Vincristine 1.5 mg/m2/dose Day 1,8 and 15; Doxorubicin 30 mg/m2/dose Day 1 and 2; (Dexrazoxane : 300 mg/m2/dose Day 1 and 2, where is available)
  Other Names: C5VD Group C
  Arms: Group C
Procedure: Biopsy — Tumors are deemed unresectable at diagnosis.
  Arms: Group B; Group C; Group D
Procedure: Resection or transplant — Ideal timing to resect of the primary tumors or transplant if if excellent response achieved at 1st or 2nd evaluation timepoint. But surgery timing is not mandated. Irrespective of the timing of surgery, patients should complete all planned protocol cycles of chemotherapy (including post transplantation). If surgical resection of the primary tumor is delayed until the end of therapy, no further post-operative chemotherapy should be given.
  Arms: Group B; Group C; Group D
Procedure: Resection of pulmonary nodules — Resection of pulmonary nodules should be considered in Group D2, patients at any cycle if continuing to respond to consolidation therapy.
  Arms: Group D
Drug: mono CDDP- Group B — Cisplatin 80 mg/m2/dose Day 1. All patients in Group B (2 arms) will receive 6 cycles of mono cisplatin chemotherapy. Each cycle lasts 2 weeks (14 days).
  Arms: Group B
Drug: Block 1 to 3 (Cisplatin, Doxorubicin) Group D — Block 1 and 2: Cisplatin 70 mg/m2/dose Day1, 8 and 15; Doxorubicin 30 mg/m2/dose, Day 8 and 9; (Dexrazoxane: 300 mg/m2/dose Day 1 and 2, where is available); Block 3: Cisplatin 70 mg/m2/dose Day1and 8; Doxorubicin 30 mg/m2/dose Day 8 and 9; (Dexrazoxane BSA ≥ 0.6 m2/dose: 300 mg/m2/dose Day 8 and 9, where is available) All patients in Group D will receive 3 blocks in induction, followed by consolidation therapy. Block 1 and 2 last 28 days. Block 3 is 21 cycles.
  Arms: Group D
Drug: Consolidation (Carboplatin, Doxorubicin) -Group D1 — Following Block 1-3 of induction therapy, Group D1 patients will receive 3 cycles of Carboplatin + Doxorubicin consolidation therapy. Each cycle lasts 3 weeks (21 days). Carboplatin 500 mg/m2/dose Day 1; Doxorubicin 20 mg/m2/dose Day 1 and 2; (Dexrazoxane: 200 mg/m2/dose Day 1 and 2, where is available).
  Other Names: Group D1 CD
  Arms: Group D
Drug: Consolidation (Carboplatin +Doxorubicin/Vincristine + Irinotecan)-Group D2 — Following Block 1-3 of induction therapy, patients in Group D2, will receive 6 cycles of consolidation chemotherapy with Carboplatin + Doxorubicin in Cycles 1, 3, and 5 alternating with Vincristine + irinotecan in Cycles 2, 4, and 6. One cycle of therapy lasts 3 weeks (21 days). Cycle 1, 3 and 5: Carboplatin 500 mg/m2/dose Day 1; Doxorubicin 20 mg/m2/dose Day 1 and 2; (Dexrazoxane: 200 mg/m2/dose Day 1 and 2, where is available).
  Cycle 2, 4 and 6: Vincristine 1.5 mg/m2/dose, Day 1 and 8; Irinotecan 50 mg/m2/dose, Day 1 to 5;
  Other Names: Group D2 CD/VI
  Arms: Group D

SUMMARY:
A Phase 3 multi-institutional study for treatment of children with newly diagnosed hepatoblastoma using a modified Paediatric Hepatic International Tumour Trial (PHITT) strategy incorporating a randomized assessment of sodium thiosulfate as auditory protection for children with localized disease, and response adapted therapy for patients with metastatic disease

DETAILED DESCRIPTION:
Primary aims:

1. Localized Disease: Groups B and C: To evaluate and validate the efficacy of sodium thiosulfate (STS) to reduce the hearing impairment caused by a cisplatin monotherapy in non-metastatic patients without adverse features (localized PRETEXT I-III tumors without positive VPEFR annotation factors) (Group B - treated with cisplatin mono-therapy) or with adverse features (localized PRETEXT I-III tumors with positive VPEFR annotation factors) (Group C - treated with regimen C5VD)
2. Metastatic Disease: Group D: To determine the 3-year Event-free survival (EFS) in patients with metastatic disease treated with International Society of Paediatric Oncology (SIOPEL 4) induction therapy followed by response adapted consolidation therapy.
3. To determine the 3-year EFS in patients with HB whose tumor is completely resected at diagnosis (Group A) and either receive no adjuvant chemotherapy (Group A1, completely resected well differentiated fetal (WDF) histology HB) or 2 cycles of standard dose cisplatin monotherapy (Group A2, completely resected non-well differentiated fetal histology HB)

Secondary aims:

1. To determine any impact of STS on chemotherapy response and survival in children with localized hepatoblastoma
2. To assess the feasibility of complete resection after 2 cycles of interval compressed lower dose cisplatin monotherapy (80 mg/m2/cycle) in non-metastatic patients and without adverse features
3. To assess the feasibility of complete resection after 2 cycles of C5VD in non-metastatic patients with adverse features.5. To determine the adherence to PRETEXT and Post-treatment extent of disease (POSTTEXT) based surgical guidelines
4. To determine the prognostic relevance in HB of a "small cell undifferentiated", tumor component, percentage of tumor necrosis in post chemotherapy specimens, and the relevance of a positive microscopic margin in resected HB specimens.
5. To determine the concordance between institutional, regional expert panel (prospective) and international expert panel (retrospective) review assessment of PRETEXT and POSTTEXT stage, and correlate with outcome variables.
6. To prospectively collect patient HB tumor, peripheral blood and urine specimens, for translational biology studies.

ELIGIBILITY:
Inclusion Criteria:

* Performance Level Patients must have a performance status corresponding to ECOG scores 0, 1, or 2. Use Karnofsky for patients >16 years of age and Lansky for patients ≤16 years of age.
* Diagnosis Patients must be newly diagnosed with histologically-proven primary pediatric HB
* Emergent Treatment for HB In emergency situation when a patient meets all other eligibility criteria and has had baseline required observations, but is too ill to undergo a biopsy safely, the patient may be enrolled without a biopsy.
* Prior Therapy Patients may have had surgical resection of the hepatic malignancy prior to enrollment. All other anti-cancer therapy for the current liver lesion is prohibited.
* Organ Function Requirements

I) Adequate renal function defined as:

Creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) ≥ 70 mL/min/1.73 m2

II) Adequate liver function defined as:

Total bilirubin ≤ 5 x upper limit of normal (ULN) for age, and Aspartate aminotransferase (AST) or Alanine transaminase (ALT) < 10 x upper limit of normal (ULN) for age.

III) Adequate pulmonary function defined as:

Normal pulmonary function tests (including DLCO) if there is clinical indication for determination (e.g. dyspnea at rest, known requirement for supplemental oxygen)

Exclusion Criteria:

* Prior chemotherapy or tumor directed therapy expect for surgical resection of the hepatic malignancy (i.e. radiation therapy, biologic agents, local therapy (embolization, radiofrequency ablation, and laser)). Therefore, patients with a pre-disposition syndrome who have a prior malignancy are not eligible.
* Patients who are currently receiving another investigational drug.
* Patients who are currently receiving other anticancer agents.
* Patients with uncontrolled infection.
* Patients who previously received a solid organ transplant.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Audiogram | From diagnosis through study completion, an average of 1 year
  The grade (from 0 to 4, higher scores mean a worse outcome) of audiograms evaluated by Boston Grading Scale for Ototoxicity.To evaluate and validate the efficacy of sodium thiosulfate (STS) to reduce the hearing impairment caused by a cisplatin monotherapy in non- metastatic patients without adverse features (localized PRETEXT I-III tumors without positive VPEFR annotation factors) (Group B - treated with cisplatin mono-therapy) or with adverse features (localized PRETEXT I-III tumors with positive VPEFR annotation factors) (Group C - treated with regimen C5VD).
3 -year Event-free survival (EFS) | UP to 3years
  Calculated from the time of randomisation to the first of the following events: progression, relapse, secondary malignancy or death.

SECONDARY OUTCOMES:
Treatment-related adverse events | UP to 3years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0
Response to chemotherapy | UP to 3years
  Complete response (CR):
  no evidence of disease and normal serum AFP value (for age).
  Partial response (PR):
  any tumour volume shrinkage associated with a decreasing serum AFP value, > 1 log below the original measurement.
  Stable disease (SD):
  no tumour volume change and no change, or < 1 log fall of the serum AFP concentration.
  Progressive disease (PD):
  unequivocal increase in 1 or more dimensions and/or any unequivocal increase of the serum AFP concentration (three successive 1-2 weekly determinations) even without clinical (physical and/or radiological) evidence of tumour re-growth.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, SAP and ICF were shared before study initiation. Patient data and the information about the process of the study will be shared within the 3 participants annually after enrollment patients.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared within the 3 hospital every 12 months after enrollment of patients.
Access Criteria: Scheduled meeting and paper transferring.

REFERENCES:
- [Background] Brock PR, Maibach R, Childs M, Rajput K, Roebuck D, Sullivan MJ, Laithier V, Ronghe M, Dall'Igna P, Hiyama E, Brichard B, Skeen J, Mateos ME, Capra M, Rangaswami AA, Ansari M, Rechnitzer C, Veal GJ, Covezzoli A, Brugieres L, Perilongo G, Czauderna P, Morland B, Neuwelt EA. Sodium Thiosulfate for Protection from Cisplatin-Induced Hearing Loss. N Engl J Med. 2018 Jun 21;378(25):2376-2385. doi: 10.1056/NEJMoa1801109. PMID 29924955
- [Background] Freyer DR, Chen L, Krailo MD, Knight K, Villaluna D, Bliss B, Pollock BH, Ramdas J, Lange B, Van Hoff D, VanSoelen ML, Wiernikowski J, Neuwelt EA, Sung L. Effects of sodium thiosulfate versus observation on development of cisplatin-induced hearing loss in children with cancer (ACCL0431): a multicentre, randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2017 Jan;18(1):63-74. doi: 10.1016/S1470-2045(16)30625-8. Epub 2016 Dec 1. PMID 27914822
- [Background] Freyer DR, Brock P, Knight K, Reaman G, Cabral S, Robinson PD, Sung L. Interventions for cisplatin-induced hearing loss in children and adolescents with cancer. Lancet Child Adolesc Health. 2019 Aug;3(8):578-584. doi: 10.1016/S2352-4642(19)30115-4. Epub 2019 May 31. PMID 31160205
- [Background] Meyers RL, Maibach R, Hiyama E, Haberle B, Krailo M, Rangaswami A, Aronson DC, Malogolowkin MH, Perilongo G, von Schweinitz D, Ansari M, Lopez-Terrada D, Tanaka Y, Alaggio R, Leuschner I, Hishiki T, Schmid I, Watanabe K, Yoshimura K, Feng Y, Rinaldi E, Saraceno D, Derosa M, Czauderna P. Risk-stratified staging in paediatric hepatoblastoma: a unified analysis from the Children's Hepatic tumors International Collaboration. Lancet Oncol. 2017 Jan;18(1):122-131. doi: 10.1016/S1470-2045(16)30598-8. Epub 2016 Nov 22. PMID 27884679
- [Background] Brock PR, Knight KR, Freyer DR, Campbell KC, Steyger PS, Blakley BW, Rassekh SR, Chang KW, Fligor BJ, Rajput K, Sullivan M, Neuwelt EA. Platinum-induced ototoxicity in children: a consensus review on mechanisms, predisposition, and protection, including a new International Society of Pediatric Oncology Boston ototoxicity scale. J Clin Oncol. 2012 Jul 1;30(19):2408-17. doi: 10.1200/JCO.2011.39.1110. Epub 2012 Apr 30. PMID 22547603
- [Background] Zsiros J, Brugieres L, Brock P, Roebuck D, Maibach R, Zimmermann A, Childs M, Pariente D, Laithier V, Otte JB, Branchereau S, Aronson D, Rangaswami A, Ronghe M, Casanova M, Sullivan M, Morland B, Czauderna P, Perilongo G; International Childhood Liver Tumours Strategy Group (SIOPEL). Dose-dense cisplatin-based chemotherapy and surgery for children with high-risk hepatoblastoma (SIOPEL-4): a prospective, single-arm, feasibility study. Lancet Oncol. 2013 Aug;14(9):834-42. doi: 10.1016/S1470-2045(13)70272-9. Epub 2013 Jul 4. PMID 23831416